CLINICAL TRIAL: NCT03672838
Title: A Single Center Pilot Study to Assess the Intra-observer Reliability of Measuring Muscle Strength Using a Hand Held Dynamometer in Children and Adults With Neurofibromatosis Type 1 (NF1) and Type 2 (NF2).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-00831
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Neurofibromatosis 1 and 2 (NF1 and NF2)
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibromatosis 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Active Comparator): Patients with NF1
  Interventions: Behavioral: hand-held dynamometer
- Cohort 2 (Active Comparator): Patients with NF2
  Interventions: Behavioral: hand-held dynamometer

INTERVENTIONS:
Behavioral: hand-held dynamometer — Strength of one weak muscle group and of the biceps of the dominant arm will be measured using a hand-held dynamometer. An average of three readings will be used as one observation. Three observations per patient will be obtained on one day with a minimum of 15 minute rest period between each observation.

SUMMARY:
Patients with clinically confirmed neurofibromatosis type 1 (NF1) or neurofibromatosis type 2 (NF2) or a known neurofibromatosis (NF) mutation aged 5 years and above will be eligible to participate and will be recruited from the neurofibromatosis clinic. Given the need for identifying measures that can reliably and sensitively measure focal muscle weakness and allow for measuring muscle strength as a functional outcome in therapeutic clinical trials in NF, this pilot study will assess the reliability of measuring muscle strength in NF1 and NF2 using a hand-held dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* For cohort 1:

  * Patients must have clinically confirmed NF1 using the NIH consensus criteria or a known NF1 mutation
  * Ages 5 years and above
  * < 5/5 strength on Manual Muscle Testing (MMT) testing in at least one muscle group tested on the day of enrollment
  * Able to follow instructions and cooperate with exam to assess strength
* For Cohort 2

  * Patients must have clinically (NIH or Manchester criteria) or genetically confirmed diagnosis of NF2
  * Ages 5 years and above
  * < 5/5 strength on MMT testing in at least one muscle group tested on the day of enrollment
  * Able to follow instructions and cooperate with exam to assess strength

Exclusion Criteria:

* No orthopedic procedure or other major surgery that could influence extremity strength in past 6 months
* No tibial dysplasia

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Intra-class correlation coefficient of strength measurement in the clinically identified weak muscle | 1 day
  A sample size of 20 subjects with three observations per subject achieves 90% power to detect an intraclass correlation of 0.91 under the alternative hypothesis when the intraclass correlation under the null hypothesis is 0.75 using an F-test with a significance level of 0.05.

SECONDARY OUTCOMES:
Intra-class correlation coefficient of strength measurement in the dominant biceps | 1 day
  A sample size of 20 subjects with three observations per subject achieves 90% power to detect an intraclass correlation of 0.91 under the alternative hypothesis when the intraclass correlation under the null hypothesis is 0.75 using an F-test with a significance level of 0.05.
standard error of measurement of measuring strength in the weak muscles | 1 day
standard error of measurement of measuring strength in the dominant biceps muscle | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Kaleb H Yohay, MD, Principal Investigator — New York School of Medicine
Locations (1):
- New York School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for patients who consent for their data to be shared for future research.
  The data will be made available: Requests should be directed to xxx@yyy. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose will have access to the data.